CLINICAL TRIAL: NCT02226419
Title: Fat and Carbohydrate Metabolism During Exercise, With and Without L-carnitine Supplementation in Patients With Carnitine Transporter Deficiency
Brief Title: Fat and Sugar Metabolism During Exercise, With and Without L-carnitine in Patients With Carnitine Transporter Deficiency
Acronym: CTD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Lindhardt Madsen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Karen Lindhardt Madsen, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1-2012-130
Record Dates: First submitted 2013-08-05; First posted 2014-08-27 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Carnitine Transporter, Plasma-membrane, Deficiency of
Keywords: Fatty acid oxidation disorder; Primary carnitine deficiency; Exercise; L-carnitine treatment; Stable isotopes; Carnitine transporter deficiency
MeSH Terms: conditions — Systemic carnitine deficiency; Motor Activity | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Break in L-carnitine treatment (Experimental): Patients do not take their L-carnitine (Levocarnitine) treatment for 2-4 days until plasma carnitine and acylcarnitine have fallen. While patients abstain from taking the treatment, they are admitted for cardiac telemetry monitoring.
  Interventions: Dietary Supplement: Break in L-carnitine treatment

INTERVENTIONS:
Dietary Supplement: Break in L-carnitine treatment — Levocarnitine oral tablet supplement at individual doses
  Other Names: Levocarnitine

SUMMARY:
The investigators wish to investigate fat and sugar metabolism during exercise with and without L-carnitine supplementation in patients with carnitine transporter deficiency (CTD).

Patients with CTD have low plasma- and muscle concentrations of carnitine, which is believed to lead to an impaired fat oxidation. Presently there is no cure available for these patients, but daily intake of L-carnitine has been shown to limit the amount of symptoms. Little is known about the metabolism during exercise and the pathophysiological mechanisms causing the symptoms.

Studying the fat and sugar metabolism in CTD patients will contribute to the understanding of the role of the carnitine transporter in the development of symptoms in these patients. Furthermore, knowledge about the fat and sugar metabolism in these patients can increase the understanding of the role of the carnitine transporter in the metabolism healthy persons.

The investigators have included 8 patients with genetically verified CTD in the study and a group of 10 age- and sex-matched controls. Subjects will perform a 1h cycling test, exercising at a moderate intensity. By measuring the expiration of carbon dioxide (CO2) and consumption of oxygen (O2), the investigators can determine the total fatty acid and carbohydrate oxidation during cycling. At the same time the investigators will measure the patients' whole body palmitate (fat) and glucose (sugar) oxidation rates using stable isotope technique.

The patient group will repeat the cycling test after 4 days without taking their usual L-carnitine treatment. During the treatment break, patients will be admitted to be continuously monitored for heart rhythm disturbances, which is a known but rarely occurring complication to untreated CTD.

Since the patients have a defect in their fat metabolism, the investigators expect to find that they have a reduced ability to burn fat, which is the major source of energy during low intensity exercise. It is therefore likely, that the CTD patients will benefit from adjustments in their daily diet, whenever they have to perform physically. By learning about the metabolism of different dietary substances, fat and sugar, these studies can help to improve the treatment in terms of dietary recommendations for CTD patients. This will have a direct impact on the daily life of the patients.

DETAILED DESCRIPTION:
8 Patients with verified CTD have been included

* All patients have performed an incremental load exercise test to exhaustion on a cycle ergometer to determine maximal oxygen comsumption rate (VO2 max)
* One-hour exercise test: Measurement of the total fat and sugar oxidation rates during exercise using stable isotope tracers.

Subjects arrive at the laboratory after 3-9 hours fasting. One IV-catheter is inserted in the cubital vein in one arm and another in a peripheral vein in the other hand. The stable isotope tracers will be given in the cubital vein as a constant infusion of solutions of:

* [U-13C]-palmitate (0.0026 mg x kg-1 x min-1, after a priming bolus of 0.085 mg x kg-1 NaH13CO3)
* [1,1,2,3,3-2H5]-glycerol (0.0049 mg x kg-1 x min-1 )
* [6.6-2H2]-glucose (0.0728 mg x kg-1 x min-1 ) 5 days before the study, subjects must avoid eating food containing corn. Corn contains larger amounts of C13, which we use as a tracer, and can therefore disturb the measurements.

For two hours the subjects rest while receiving the infusions until the tracers have distributed in the body and reached a steady state. After the rest, the subjects exercise on the cycle-ergometer until exhaustion or for a maximum of 1 hour at an intensity that corresponds to 60-70% of VO2max.

Every other minute during exercise, the heart rate is recorded and the subject evaluates his/her degree of exertion (Rate of Perceived Exertion, RPE) on a Borg scale.

Blood and breath samples:

From 20 minutes before exercise until the end of exercise, blood samples are drawn through the IV-catheter in the hand vein (10-12 mL per sample) and samples of the expired breath are collected in a Douglas bag (Hans Rudolph inc.) every ten minutes. The breath is transferred into Vaccutainer-glas for analysis of 13CO2 -enrichment (10 mL). The plasma samples are anayzed for concentrations of hormones, metabolites, carnitine and acyl-carnitines.

Muscle biopsy:

On this day a muscle biopsy is taken from the vastus lateralis of the thigh to measure the intramuscular concentrations of carnitine and acylcarnitines.

* Wash-out period: For 4 days patients were admitted for telemetric cardiac monitoring while they pause their daily oral L-carnitine treatment.
* After the washout period, patients repeat the one-hour exercise test with the stable isotope tracers. Also the muscle biopsy for intramuscular carnitine and acyl-carnitine concentrations are repeated-

TRACERS In this study we will use infusions of stable isotopes incorporated into metabolites as tracers of whole body metabolism. We will use small amounts of fat (palmitate and glycerol) and sugar (glucose) labelled with stable isotopes of carbon (13C) and hydrogen (2H). The palmitate and glycerol tracers (98 % enriched, Cambrigde Isotope Laboratories, Andover, MA, USA) will be dissolved in sterile water and infused through a bacterial filter into human serum albumin. The glucose tracer (99 % enriched, Cambrigde Isotope Laboratories, Andover, MA, USA) will be dissolved and injected into a solution of 0.9% saline (NaCl) through a bacterial filter as well.

These tracers are naturally occurring in food (e.g. in corn) and in the human body. They are harmless and will be handled and given to the subjects under sterile conditions.

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis of CTD

Exclusion Criteria:

* Other conditions or diseases that may compromise the outcome of the study
* Pregnancy or lactation
* Inability to cooperate carrying out the experiments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The whole body palmitate and carbohydrate oxidation rate in CTD patients during exercise | With and without L-carnitine treatment
  The whole body palmitate and carbohydrate oxidation will be assessed during 1h exercise test performed on a cycle-ergometer using stable isotope technique combined with indirect calorimetry.

SECONDARY OUTCOMES:
The maximal oxidative capacity (VO2max) as an indicator of exercise tolerance and performance in CTD patients | During a 15 min incremental intensity exercise test and during a 1h moderate intensity cycling test

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Madsen, MD, Principal Investigator — Neuromuscular Research Unit, Rigshospitalet

REFERENCES:
- [Derived] Madsen KL, Preisler N, Rasmussen J, Hedermann G, Olesen JH, Lund AM, Vissing J. L-Carnitine Improves Skeletal Muscle Fat Oxidation in Primary Carnitine Deficiency. J Clin Endocrinol Metab. 2018 Dec 1;103(12):4580-4588. doi: 10.1210/jc.2018-00953. PMID 30219858